CLINICAL TRIAL: NCT01624415
Title: Subjective Image Quality in Stereoscopic Image Modifications
Acronym: Stereopsis
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, MD, assco. Prof., Medical University of Vienna
Other Study IDs: OPHT - 190312
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Stereoscopic Vision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Humans attain binocular vision from the two retinal images of both eyes through a series of sensory and motor processes that culminate in the perception of stereoscopic depth. Looking at a scene creates two slightly different images on the retinas which is due to the eyes' different positions on the head. This so called binocular disparity provides information to calculate depth and therefore enables stereopsis. Physiologically the two retinal images are superimposed and merge into one stereoscopic image.

If one image is presented to one eye in an experimental setting, and a completely different image is presented to the other eye, the investigators visual system, analogous to diplopic vision, is not able to fuse these image stimuli. Instead, a phenomenon called binocular rivalry occurs. Here, both images are seen alternating and the brain can switch back and forth between these images.

The aim of the present study is to investigate the effects of objective changes to image quality on the investigators subjective stereoscopic perception. This psychophysiological testing is done by looking at different images and thereafter by subjective grading of the image quality.

The investigators hypothesize that overlapping image modifications occurring in both eyes are detected immediately, but changes, that are rotated by 90 degrees against each other, should be suppressed and result in one stereoscopic image, reduced in image quality. Whether this also accounts for more detailed images, such as reading cards, is questionable.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years, nonsmokers
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, emmetropia or ≤ 1 diopter

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except oral contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants will be selected by the Department of Clinical Pharmacology healthy subjects, male and female, 18-35 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria